CLINICAL TRIAL: NCT04143399
Title: Holmium Laser Enucleation vs Bipolar Resection of a Large Volume BPH: a Randomised Controlled Study
Brief Title: HoLEP vs BPRP of a Large Volume BPH: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSheemy, Professor of Urology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 62513
Record Dates: First submitted 2019-10-26; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: BPH With Urinary Obstruction; Male
Keywords: BPH; enucleation; Large Prostate; LUTS; IPSS; quality of life

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- holmium laser enucleation of the prostate (Active Comparator): holmium laser enucleation of the prostate (HoLEP)
  Interventions: Procedure: holmium laser enucleation of the prostate
- bipolar resection of the prostate (Active Comparator): bipolar resection of the prostate (BPEP)
  Interventions: Procedure: Bipolar resection of the prostate

INTERVENTIONS:
Procedure: holmium laser enucleation of the prostate — cystoscopic transurethral enucleation of the prostate using Holmium laser (Versa pulse 100W; Lumenis; Germany)
  Other Names: HoLEP
  Arms: holmium laser enucleation of the prostate
Procedure: Bipolar resection of the prostate — cystoscopic transurethral resection of the prostate using bipolar energy
  Other Names: BPRP
  Arms: bipolar resection of the prostate

SUMMARY:
To compare bipolar resection versus holmium laser enucleation for management of large BPH.

DETAILED DESCRIPTION:
To compare safety and efficacy of bipolar resection (BPRP) versus holmium laser enucleation (HoLEP) for management of large BPH (> 75 gm).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from LUTS secondary to infravesical obstruction from BPH
* failed medical treatment
* International Prostate Symptom Score (IPSS) > 13
* a peak urinary flow rate (Qmax) < 15 ml/sec
* a prostate size ≥ 75 gm

Exclusion Criteria:

* presence of a urethral stricture
* neurological disorder
* bladder cancer
* prostate cancer
* previous history of bladder neck surgery or TURP

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-02-14 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
hemoglobin drop postoperatively (gm/dL) | Immediate postoperatively
  difference in hemoglobin concentration postoperatively vs preoperatively
operative duration in minutes | during surgery
  operative duration
Hospital stay in days | immediately after surgery
  Hospital stay

SECONDARY OUTCOMES:
complications (%) | Two years
  intraoperative and postoperative complications including blood transfusion, capsular perforation, irritative symptoms, SUI, urethral stricture, bladder neck contracture, urinary retention.
urine flow | Two years
  Qmax (ml/s),
post-voiding residual urine | Two years
  postvoiding residual urine (ml)
International prostate symptom score (IPSS) | Two years
  an international commonly used score ranging from 0 - 35 (the worst is 35) evaluating voiding and storage urinary symptoms using 7 questions each one is scored from 0 to 5 according to severity of symptom
Quality of life (QoL) | Two years
  section of International prostate symptom score (IPSS) one question scored from 0 up to 6 (6 is worst)
Catheter duration | immediate postoperatively
  Catheter duration in hours

CONTACTS AND LOCATIONS:
Overall Officials: enmar I Habib, Study Director — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habib EI, ElSheemy MS, Hossam A, Morsy S, Hussein HA, Abdelaziz AY, Abdelazim MS, Fathy H. Holmium Laser Enucleation Versus Bipolar Plasmakinetic Resection for Management of Lower Urinary Tract Symptoms in Patients with Large-Volume Benign Prostatic Hyperplasia: Randomized-Controlled Trial. J Endourol. 2021 Feb;35(2):171-179. doi: 10.1089/end.2020.0636. Epub 2020 Oct 29. PMID 32842769